CLINICAL TRIAL: NCT01924923
Title: New Biopsy Technique for Uveal Melanoma
Status: Completed | Type: Observational
Sponsor: Greater Houston Retina Research (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Amy C Schefler, MD, Director of Ophthalmic Oncology, Greater Houston Retina Research
Other Study IDs: NBT-01
Record Dates: First submitted 2013-08-13; First posted 2013-08-19 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Uveal Melanoma
Keywords: uveal melanoma; biopsy; enucleation; ocular cancer
MeSH Terms: conditions — Uveal Melanoma; Eye Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The eye will be enucleated and histopathologic sections of the sclera will be examined for extra scleral extension of cells. After the tissues are examined, they will be stored in the ocular histopathology lab for 10 years.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Uveal Melanoma: Scheduled for enucleation surgery

SUMMARY:
This pilot study intends to investigate a new biopsy technique that will decrease the incidence of tumor cells in the biopsy tract.

DETAILED DESCRIPTION:
Uveal melanoma is the most common primary malignancy of the eye and is one of the few fatal diseases that are detected initially through an eye examination. For many years, clinical decision-making regarding which patient with uveal melanoma required treatment has been based solely on clinical features observed at the time of diagnosis. These features include: tumor size as measured by ultrasound, associated subretinal fluid, presence of orange lipofuscin pigment, lack of drusen, posterior location, and ciliary body involvement. All of these clinical features have been demonstrated to be associated with tumor growth which is associated with the eventual development of metastases. However, these clinical features are not adequately sensitive or specific enough to predict which patients will develop metastases.

More recently, researchers studying the genomics of uveal melanoma have focused on identifying genetic abnormalities present in tumor tissue in order to characterize these lesions more fully. Several landmark papers over the past 15 years have reported cytogenic and genomic abnormalities in uveal melanoma tumor tissue that are associated with a poorer prognosis. Although rare, there have been at least five cases in which patients undergoing biopsy of these lesions have developed extraocular spread of melanoma from the biopsy sites. With this new technique, the possible rate of extraocular spread should be lower, making the biopsy a safer technique than what is currently in practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with uveal melanoma
* Scheduled for enucleation surgery

Exclusion Criteria:

* Patients under 21 years old
* Patients unable to undergo surgery
* Patients with known metastatic uveal melanoma or other cancer.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 21, diagnosed with uveal melanoma and scheduled to undergo enucleation surgery. No known metastatis.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects with melanotic cells present at biopsy needle site | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Amy C. Schefler, MD, Principal Investigator — Retina Consultants Houston
Locations (1):
- Retina Consultants of Houston, Houston, Texas, United States

REFERENCES:
- [Background] The Collaborative Ocular Melanoma Study (COMS) randomized trial of pre-enucleation radiation of large choroidal melanoma III: local complications and observations following enucleation COMS report no. 11. Am J Ophthalmol. 1998 Sep;126(3):362-72. doi: 10.1016/s0002-9394(98)00091-9. PMID 9744369
- [Background] The Collaborative Ocular Melanoma Study (COMS) randomized trial of pre-enucleation radiation of large choroidal melanoma II: initial mortality findings. COMS report no. 10. Am J Ophthalmol. 1998 Jun;125(6):779-96. doi: 10.1016/s0002-9394(98)00039-7. PMID 9645716
- [Background] Schyberg E. Fine needle biopsy of orbital tumours [proceedings]. Acta Ophthalmol Suppl. 1975;(125):11. doi: 10.1111/j.1755-3768.1975.tb01202.x. No abstract available. PMID 184645
- [Background] Jakobiec FA, Coleman DJ, Chattock A, Smith M. Ultrasonically guided needle biopsy and cytologic diagnosis of solid intraocular tumors. Ophthalmology. 1979 Sep;86(9):1662-81. doi: 10.1016/s0161-6420(79)35349-0. PMID 551354
- [Background] Caminal JM, Sanz S, Carreras M, Catala I, Arruga J, Roca G. Epibulbar seeding at the site of a transvitreal fine-needle aspiration biopsy. Arch Ophthalmol. 2006 Apr;124(4):587-9. doi: 10.1001/archopht.124.4.587. No abstract available. PMID 16606890
- [Background] Glasgow BJ, Brown HH, Zargoza AM, Foos RY. Quantitation of tumor seeding from fine needle aspiration of ocular melanomas. Am J Ophthalmol. 1988 May 15;105(5):538-46. doi: 10.1016/0002-9394(88)90248-6. PMID 3369520
- [Background] Karcioglu ZA, Gordon RA, Karcioglu GL. Tumor seeding in ocular fine needle aspiration biopsy. Ophthalmology. 1985 Dec;92(12):1763-7. doi: 10.1016/s0161-6420(85)34105-2. PMID 4088631
- [Background] Engzell U, Esposti PL, Rubio C, Sigurdson A, Zajicek J. Investigation on tumour spread in connection with aspiration biopsy. Acta Radiol Ther Phys Biol. 1971 Aug;10(4):385-98. doi: 10.3109/02841867109130784. No abstract available. PMID 4329702
- [Background] SNELL AC Jr. Heterotransplantation of tumors into various regions of the guinea-pig eye. Am J Ophthalmol. 1951 May;34(5 1):733-8. doi: 10.1016/0002-9394(51)92285-4. No abstract available. PMID 14829489
- [Background] Shields JA, Shields CL, Ehya H, Eagle RC Jr, De Potter P. Fine-needle aspiration biopsy of suspected intraocular tumors. The 1992 Urwick Lecture. Ophthalmology. 1993 Nov;100(11):1677-84. doi: 10.1016/s0161-6420(93)31418-1. PMID 8233394
- [Background] Schefler AC, Gologorsky D, Marr BP, Shields CL, Zeolite I, Abramson DH. Extraocular extension of uveal melanoma after fine-needle aspiration, vitrectomy, and open biopsy. JAMA Ophthalmol. 2013 Sep;131(9):1220-4. doi: 10.1001/jamaophthalmol.2013.2506. PMID 24030334